CLINICAL TRIAL: NCT04064814
Title: Evaluation of Efficacy and Safety of add-on Alpha-lipoic Acid on Migraine Prophylaxis in Adolescent Population: A Randomized Controlled Trial
Brief Title: Evaluation of Efficacy and Safety of add-on Alpha-lipoic Acid on Migraine Prophylaxis in Adolescent Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Assistant professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIIMSBBSR/PGThesis/2019-20/15
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Adolescent Migraine
Keywords: Adolescent Migraine; Flunarizine; Alpha Lipoic Acid; Thiol Level; Calcitonin gene regulated peptide
MeSH Terms: interventions — Flunarizine; Thioctic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, open Label , active controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flunarizine (Active Comparator): flunarizine will be prescribed at a dose of 5mg once daily , orally for 12 weeks
  Interventions: Drug: Flunarizine 5mg
- Alpha Lipoic Acid (Experimental): Alpha Lipoic Acid will be prescribed at a dose of 300mg once daily,orally for 12 weeks
  Interventions: Drug: Flunarizine 5mg; Drug: Alpha lipoic acid 300mg

INTERVENTIONS:
Drug: Flunarizine 5mg — Flunarizine 5mg once daily,orally for 12 weeks
Drug: Alpha lipoic acid 300mg — Alpha lipoic acid 300mg ,once daily ,orally for 12 weeks
  Arms: Alpha Lipoic Acid

SUMMARY:
Migraine causes a substantial impact on the physical and mental health of a child and it is a major cause for time-off school leading to impaired academic performance. Therefore prophylactic treatment is suggested for adolescents with frequent or disabling migraine, aiming at improving the function, quality of life and reducing disability.

The most commonly used non-pharmacological agents for the prophylactic management of migraine in adolescents are nutraceuticals. Amongst all nutraceuticals, most commonly used agents for prophylaxis are coenzyme Q10, magnesium, riboﬂavin, feverfew and butterbur .

Alpha-lipoic acid (ALA) or 6,8-thioctic acid, is an endogenous molecule which functions as an important co-factor for various enzyme complexes in mitochondria and plays an important role in energy metabolism.ALA is a nutraceutical agent which also has neuroprotective and anti-inﬂammatory effects. It has been proved that the thiol level remains low in migraine patients.

However, only one study has been done by Ali et al in the pediatric population where the combination of ALA and topiramate has shown promising results but the study result is not generalizable due to its inherent limitations.

So, the study has been planned with an aim to evaluate the efficacy and safety of ALA as add-on therapy with flunarizine in the adolescent age group

DETAILED DESCRIPTION:
Migraine causes a substantial impact on the physical and mental health of a child and it is a major cause for time-off school leading to impaired academic performance. Therefore prophylactic treatment is suggested for adolescents with frequent or disabling migraine, aiming at improving the function, quality of life and reducing disability. Pharmacological agents commonly used for migraine prophylaxis in adolescents are topiramate, cyproheptadine, amitriptyline, valproate, propranolol and flunarizine. These preventive medications are effective first-line treatment but the associated adverse effects have limited their use amongst the adolescent population. In this clinical scenario nutraceuticals may be an alternative option.

The most commonly used non-pharmacological agents for the prophylactic management of migraine in adolescents are nutraceuticals. Amongst all nutraceuticals, most commonly used agents for prophylaxis are coenzyme Q10, magnesium, riboﬂavin, feverfew and butterbur . Despite being largely used for prophylaxis of adolescent migraine, sufficient evidences are lacking which support the safety and efficacy of these agents. The findings from the previous studies on riboflavin and coenzyme Q10 are conflicting and inconclusive. Thus there is a need for a clinically effective nutraceutical in migraine prophylaxis.

Alpha-lipoic acid (ALA) or 6,8-thioctic acid, is an endogenous molecule which functions as an important co-factor for various enzyme complexes in mitochondria and plays an important role in energy metabolism. ALA is a nutraceutical agent which also has neuroprotective and anti-inﬂammatory effects. It has been proved that the thiol level remains low in migraine patients. In some recent studies, ALA has been found to be beneficial in migraine prophylaxis in adults. However, only one study has been done by Ali et al in the pediatric population where the combination of ALA and topiramate has shown promising results but the study result is not generalizable due to its inherent limitations.

From the literature search, it is evident that there is a lack of data on the efficacy and safety of ALA as a prophylactic agent in migraine. So, the study has been planned with an aim to evaluate the efficacy and safety of ALA as add-on therapy with flunarizine in the adolescent age group. The choice of flunarizine as standard prophylactic therapy in the present study is supported by the fact that flunarizine is efficacious and safer in the adolescent population due to its fewer adverse effects in comparison to topiramate and propranolol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "15 or more headache days per month with at least 8 days having migraine features for at least 3 months (according to the criteria of the International Classification of Headache Disorders, 3rd edition [beta version], or ICHD-3 beta)."
* Adolescent migraineurs aged 10 to 19 years of age of either sex.
* Patients who have not taken any prophylactic treatment within the last three months before their inclusion in the study.
* Patients and/or parents have given informed written consent/assent.

Exclusion Criteria:

* Patient with headache other than migraine.
* Patients who were on corticosteroids
* Treatment with any test drugs in the preceding three months from the start of the trial.
* If there is any history of interventions or devices used for the treatment of migraine, such as transcranial magnetic stimulation and nerve blocks during the 3 months before screening.
* Any other accompanying systemic illness; abnormalities revealed on neurologic examination.
* Psychiatric disturbances, history of epilepsy , learning disabilities, head trauma or use of other drugs acting on the central nervous system, including, smoking, alcohol consumption or any illicit drug abuse

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Mean monthly migraine attack rate | 12 weeks
  Change in the mean monthly migraine attack rate from baseline after treatment with Flunarizine vs Alpha Lipoic Acid

SECONDARY OUTCOMES:
Responder rate | 12 weeks
  percentage of patients having ≥50% reduction in migraine frequency from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
The number of days with migraine headache | 12 weeks
  The number of days with migraine headache from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
The mean severity of acute attacks | 12 weeks
  The mean severity of acute attacks will be considered as severity basis where 3 will be severe and 1 will be mild attack (on a 3-point scale: 3, severe; 2, moderate; 1, mild) from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
The number of days with nausea or vomiting | 12 weeks
  The number of days with nausea or vomiting from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
The headache disability will be assessed by pedMIDAS (pediatric migraine disability assessment score) | 12 weeks
  The headache disability will be assessed by pedMIDAS (pediatric migraine disability assessment score) scoring system (denotes 0 to 10 as little to no dyability and greater than 50 as severe disability) from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
The relapse rate among the responders after stoppage of prophylactic therapy . | 12 weeks
  The relapse rate among the responders after stoppage of prophylactic therapy over the next 12 weeks.
Serum thiol levels | 12 weeks
  Serum thiol levels from baseline after treatment with Flunarizine vs Alpha Lipoic Acid
Serum CGRP | 12 weeks
  Serum CGRPlevels from baseline after treatment with Flunarizine vs Alpha Lipoic Acid

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Director — Additional Professor
Locations (1):
- AIIMS, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karsan N, Prabhakar P, Goadsby PJ. Premonitory Symptoms of Migraine in Childhood and Adolescence. Curr Pain Headache Rep. 2017 Jul;21(7):34. doi: 10.1007/s11916-017-0631-y. PMID 28647791
- [Background] Eiland LS, Jenkins LS, Durham SH. Pediatric migraine: pharmacologic agents for prophylaxis. Ann Pharmacother. 2007 Jul;41(7):1181-90. doi: 10.1345/aph.1K049. Epub 2007 Jun 5. PMID 17550953
- [Background] O'Brien HL, Kabbouche MA, Hershey AD. Treating pediatric migraine: an expert opinion. Expert Opin Pharmacother. 2012 May;13(7):959-66. doi: 10.1517/14656566.2012.677434. Epub 2012 Apr 14. PMID 22500646
- [Background] D'Onofrio F, Raimo S, Spitaleri D, Casucci G, Bussone G. Usefulness of nutraceuticals in migraine prophylaxis. Neurol Sci. 2017 May;38(Suppl 1):117-120. doi: 10.1007/s10072-017-2901-1. PMID 28527067
- [Background] Wang J, Tang J, Zhou X, Xia Q. Physicochemical characterization, identification and improved photo-stability of alpha-lipoic acid-loaded nanostructured lipid carrier. Drug Dev Ind Pharm. 2014 Feb;40(2):201-10. doi: 10.3109/03639045.2012.753901. Epub 2013 Jan 22. PMID 23336811
- [Background] Magis D, Ambrosini A, Sandor P, Jacquy J, Laloux P, Schoenen J. A randomized double-blind placebo-controlled trial of thioctic acid in migraine prophylaxis. Headache. 2007 Jan;47(1):52-7. doi: 10.1111/j.1526-4610.2006.00626.x. PMID 17355494
- [Background] Sorge F, De Simone R, Marano E, Nolano M, Orefice G, Carrieri P. Flunarizine in prophylaxis of childhood migraine. A double-blind, placebo-controlled, crossover study. Cephalalgia. 1988 Mar;8(1):1-6. doi: 10.1046/j.1468-2982.1988.0801001.x. PMID 3282670
- [Background] Abu-Arafeh I, Hershey AD, Diener HC, Tassorelli C; Clinical Trials Standing Committee and the Child and Adolescent Standing Committee of the International Headache Society. Guidelines of the International Headache Society for controlled trials of preventive treatment of migraine in children and adolescents, 1st edition. Cephalalgia. 2019 Jun;39(7):803-816. doi: 10.1177/0333102419842188. Epub 2019 Apr 4. PMID 30947525
- [Background] Sorge F, Marano E. Flunarizine v. placebo in childhood migraine. A double-blind study. Cephalalgia. 1985 May;5 Suppl 2:145-8. doi: 10.1177/03331024850050S227. PMID 2861907
- [Background] Kenney D, Jenkins S, Youssef P, Kotagal S. Patient Use of Complementary and Alternative Medicines in an Outpatient Pediatric Neurology Clinic. Pediatr Neurol. 2016 May;58:48-52.e7. doi: 10.1016/j.pediatrneurol.2015.11.003. Epub 2016 Jan 11. PMID 26923752
- [Derived] Puliappadamb HM, Satpathy AK, Mishra BR, Maiti R, Jena M. Evaluation of Safety and Efficacy of Add-on Alpha-Lipoic Acid on Migraine Prophylaxis in an Adolescent Population: A Randomized Controlled Trial. J Clin Pharmacol. 2023 Dec;63(12):1398-1407. doi: 10.1002/jcph.2331. Epub 2023 Aug 24. PMID 37563914